CLINICAL TRIAL: NCT03681535
Title: Phase II Study of Dose-Reduced Consolidation Radiation Therapy in Patients With Diffuse Large B-cell Lymphoma
Brief Title: Dose-Reduced Consolidation Radiation Therapy in Patients With Diffuse Large B-cell Lymphoma
Acronym: DLBCL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00100510
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: DLBCL; Reduce radiation dose
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm interventional study (Experimental): RT to 19.5-20Gy is given after 3 cycles of rituximab containing chemotherapy. RT is administered daily, 5 days per week in 1.5-2Gy fractions (treatments).
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — This phase II study will evaluate whether a reduction in the RT dose, concomitant with a decrease in the RT field size, in patients that achieve complete response and have a negative post-chemotherapy PET scan following 3 to 6 cycles of rituximab containing chemotherapy, will be associated with a low risk of in-field failure. The goal of this approach is to maintain excellent control rates while minimizing the risk of acute and late toxicity.

SUMMARY:
This phase II study will evaluate whether a reduction in radiation dose and field size will maintain a high rate of local control while minimizing the risk of acute and late toxicity .

Hypothesis: The radiation dose and treatment volume can be safely reduced from 30 Gy to 20 Gy while maintaining high rates of local control in patients who had a negative PET-CT scan following rituximab - containing chemotherapy.

DETAILED DESCRIPTION:
Chemotherapy followed by consolidation radiation therapy (RT) is a recognized treatment paradigm for DLBCL. This was initially established based on the results of 2 randomized trials conducted in the 1980s-1990s. In these studies patients were treated with 30Gy after chemotherapy (ECOG study) or 40-55Gy (SWOG study). A British National Lymphoma Investigation study showed no difference in freedom from local progression, progression-free survival or overall survival in between patients receiving 30Gy and 40-45Gy. Additionally systemic therapy for DLBCL has significantly improved since these initial studies, with the addition of rituximab to standard chemotherapy.

In a phase II study at Duke University patients with DLBCL NOS or primary mediastinal B-cell lymphoma were treated to 19.5-20Gy after achieving complete response to 4-6 cycles of chemotherapy containing rituximab. With a median follow-up of 43 months, there was only 1 local recurrence. The 5-year local control rate was 98%. Progression-free and overall survival at 5 years was 81% and 88%. Therefore, there is emerging evidence of long term favorable outcomes in localized DLBCL, while decreasing the risk of late effects by reducing the dose and volume of RT.

All participants will receive 20Gy instead of 30-36Gy after completion of at least 3 cycles of rituximab with combination chemotherapy. Participants must have a negative post chemotherapy PET-CT to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of stage I-IV diffuse large B-cell lymphoma, not otherwise specified (DLBCL NOS), as defined by the 2016 WHO classification. This would include all entities within this category including germinal center B-cell and non-germinal center B-cell subtypes and those with a double expressor phenotype. Also eligible are stage I-IV high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements and high-grade B-cell lymphoma, NOS
* Completion of at least 3 cycles of rituximab-containing, anthracycline-based combination chemotherapy
* Negative post-chemotherapy PET-CT scan or negative interim PET-CT scan performed within 2 weeks of the final cycle of chemoimmunotherapy. This is defined as a score of 1-3 on the PET Five Point (Deauville) Scale using the Modified Lugano Response Criteria for Non-Hodgkin's Lymphoma
* Absolute neutrophil count greater than 1000 and platelet count greater than 40,000
* Negative pregnancy test in women of child-bearing potential
* Signed study specific informed consent

Exclusion Criteria:

* Primary central nervous system lymphoma, primary cutaneous DLBCL, leg type. T-cell/histiocyte-rich large B-cell lymphoma, primary mediastinal (thymic) large B-cell lymphoma, or other distinct non-Hodgkin lymphomas arising from large B-cells included in the WHO classification
* Any absolute contraindications to irradiation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Local control rate | 2 years
  Local control rate of 95% measured by standard of care imaging obtained per the National Comprehensive Cancer Network guidelines

SECONDARY OUTCOMES:
Disease-free survival | 5 years
  Disease-free survival (DFS) will be defined as the time from on-study to first disease progression or death due to any cause, whichever comes first.
Overall Survival | 5 years
  Overall survival will be defines as the time from on-study to death due to any cause.
Patterns of failure | 5 years
  To examine patterns of failure we, we will tabulate the various ways that patients failed, up until the time of analysis. For example, these ways will include local only, local + distant, and distant only.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kelsey, MD, Principal Investigator — Duke Health
Locations (12):
- United States (7):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center in clinical affiliation with South Shore Hospital, Weymouth, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - University of Rochester James P. Wilmot Cancer Institute, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
- University Hospital Motol, Prague, Czechia
- University of Torino, Torino, Italy
- Juntendo University, Tokyo, Japan
- National Cancer Center of Singapore, Singapore, Singapore
- Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelsey CR, Broadwater G, James O, Chino J, Diehl L, Beaven AW, Chang C, Koontz BF, Prosnitz LR. Phase 2 Study of Dose-Reduced Consolidation Radiation Therapy in Diffuse Large B-Cell Lymphoma. Int J Radiat Oncol Biol Phys. 2019 Sep 1;105(1):96-101. doi: 10.1016/j.ijrobp.2019.02.055. Epub 2019 Mar 8. PMID 30858144